

### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Phase I/II Trial of Ipilimumab or Nivolumab with BMS-986156 and Hypofractionated Stereotactic Radiation Therapy in Patients with Advanced Solid Malignancies 2018-0419

| Study Chair: Joe Y. Chang | | |
|---|---|---|
| Participant's Name | Medical Record Number | |
| This is an informed consent and a | ithorization form for a research | etudy It includes s |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

### STUDY SUMMARY

The goal of this clinical research study is to find the highest tolerable dose of BMS-986156 plus ipilimumab or nivolumab with or without stereotactic body radiation therapy (SBRT) that can be given to patients with advanced solid tumors. The safety and effectiveness of these treatments will also be studied.

This is an investigational study. BMS-986156 is not FDA approved or commercially available. It is currently being used for research purposes only. SBRT is delivered using FDA-approved and commercially available methods. Ipilimumab is FDA approved and commercially available for the treatment of metastatic (has spread) melanoma that cannot be removed with surgery. Nivolumab is FDA approved and commercially available for the treatment of many different types of cancer.

It is considered investigational to use SBRT with ipilimumab or nivolumab and BMS-986156 to treat advanced solid tumors.

The study doctor can explain how the study drugs are designed to work.

Treatment on this study may help to control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment. If you take part in this study, you may experience side effects, some of which may be severe or fatal. You may choose not to take part in this study because it is a first in human study.

You can read a list of potential side effects below in the Possible Risks section of this consent.

If you are in Groups 1 or 2, you may receive up to 4 cycles of ipilimumab and BMS-986156 followed by 26 cycles of nivolumab with or without SBRT. If you are in Group 3, you may receive 4 cycles of nivolumab and BMS-986156 with SBRT, followed by 22 cycles of nivolumab alone.

Ipilimumab, nivolumab, and BMS-986156 will be provided at no cost to you while you are on study. You and/or your insurance provider may be responsible for the cost of SBRT while you are on study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive standard photon radiation therapy outside of this study. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

# Screening Tests

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will be performed within 14-28 days before your first cycle of treatment to help the doctor decide if you are eligible.

- You will have a physical exam.
- Blood (about 4 teaspoons) will be drawn for routine tests and to test for both hepatitis B and C as well as HIV (the AIDS virus). This routine blood draw will include a pregnancy test if you can become pregnant. To take part in this study, you must not be pregnant.
- Blood (about 2 teaspoons) will be drawn for biomarker testing (including genetic biomarkers), if the doctor thinks it is safe for this sample to be collected.
   Biomarkers are found in the blood/tissue and may be related to your reaction to the study drugs.
- Urine will be collected for routine tests.
- You will have an MRI, CT, or PET-CT scan to check the status of the disease.
- You may have a 4-dimension CT (4DCT) scan of your chest to check the status
  of the disease and to help the doctors decide what dose of SBRT you will
  receive. A 4DCT is a type of CT scan that looks at how the tumor may move
  when you are breathing. You may be asked to hold your breath for short periods
  of time during this test.
- You will have an EKG to check your heart function.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

### Study Groups

If you are found to be eligible to take part in this study, you will be assigned to 1 of 3 treatment groups based on when you join the study, the type of disease you have, and what the doctor thinks is in your best interest. The dose of study drugs you receive will depend on which treatment group you are in. The study staff will discuss this with you.

## Group 1: BMS-986156, ipilimumab, and nivolumab

In **Group 1**, you will receive ipilimumab, BMS-986156, and nivolumab. Up to 20 participants will be enrolled in Group 1 of the study. All participants will receive the same dose level of nivolumab and ipilimumab. You may receive 1 of 2 dose levels of BMS-986156. The first group of participants will receive the lowest dose level of BMS-986156. The next group will receive a higher dose of BMS-986156 than the group before it, if no intolerable side effects were seen. One (1) of these 2 doses will be selected for Group 2.

### Group 2: BMS-986156, ipilimumab, nivolumab, and SBRT

In Group 2, you will receive BMS-986156, ipilimumab, nivolumab, and SBRT. The dose of ipilimumab, nivolumab, and SBRT will not change. The dose of BMS-986156 you receive will be the dose selected in Group 1. Up to 20 participants will be enrolled in Group 2.

### Group 3: BMS-986156, nivolumab, and SBRT

In Group 3, you will receive BMS-986156, nivolumab, and SBRT. All participants will start with the same dose of study drugs. Based on the results of Groups 1 and 2 and your response to the study drugs, the dose may be changed.

Up to 60 participants will be enrolled in this study. All will take part at MD Anderson.

### Study Drug Administration

Study cycles for Group 1 and 2 is 21 days for the first 4 cycles followed by 28 days each for up to an additional 26 cycles. For Group 3, each cycle is 28 days for up to 26 cycles.

### Group 1

You will receive ipilimumab by vein over about 90 minutes and BMS-986156 by vein over about 60 minutes on Day 1 of Cycles 1-4. You will not receive ipilimumab or BMS-986156 after Cycle 4. Starting on Day 1 of Cycle 5, you will receive nivolumab by vein over about 30 minutes for up to 26 cycles.

### Group 2

You will receive ipilimumab by vein over about 90 minutes and BMS-986156 by vein over about 60 minutes on Day 1 of cycles 1 and 2. Then, on Days 29-32 or 29-40 of

the study (depending on the dose of SBRT you are receiving), you will receive SBRT. The study staff will explain how the radiation therapy is given.

After your SBRT treatment, you will receive ipilimumab and BMS-986156 on Day 1 of Cycles 3 and 4. You will not receive ipilimumab or BMS-986156 after Cycle 4. Starting on Day 1 of Cycle 5, you will receive nivolumab by vein over about 30 minutes for up to 26 cycles.

### Group 3

You will receive nivolumab by vein over about 30 minutes and BMS-986156 by vein over about 60 minutes on Day 1 of Cycle 1. You will also receive SBRT over about 30-45 minutes on Days 1-4 or 1-12 of Cycle 1. After your SBRT treatment, you will receive nivolumab and BMS-986156 by vein on Day 1 of Cycles 2-4. Starting on Day 1 of Cycle 5, you will receive nivolumab by vein over about 30 minutes for up to 22 cycles.

You will be given standard drugs to help decrease the risk of side effects and to help support your immune system. You may ask the study staff for information about how the drugs are given and their risks.

You will no longer be able to receive treatment if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after you have completed the follow-up visits.

### **Study Visits**

**Before your first dose of study drug**, you will have a core tumor biopsy and blood (about 6 teaspoons) will be drawn to check the status of the disease and for biomarker testing. To perform a core biopsy, you will be given local anesthesia and a sample of tissue is removed using a hollow core needle that has a cutting edge.

# During Week 1 of all cycles:

- You will have a physical exam.
- Blood (about 1 tablespoon) will be drawn for routine tests.

During Week 1 of Cycle 2 (Groups 1 and 3) or Week 3 of Cycle 2 (Group 2), you will have a tumor biopsy drawn for biomarker testing. Blood (about 6 teaspoons) will be drawn at this time for participants in Group 1/ Participants in Groups 2 and 3 will have this blood draw performed on the last day of radiation treatment. If the disease gets worse at any time on study, this biopsy and blood draw will be repeated.

During Week 1 of Cycle 5 (Groups 1 or 2) or Week 1 of Cycle 3 (Group 3), you will have an MRI, CT scan, and/or PET/CT scan to check the status of the disease. After that, you will have additional scans performed every 2-4 months while you are actively receiving treatment to check the status of the disease.

### Follow-Up

About 30 days after your last dose of nivolumab and then every 2-4 months after that for up to 1 year, you will come to the clinic for follow-up visits. At these visits:

- You will have a physical exam.
- Blood (about 1 tablespoon) be drawn for routine tests.
- You will have an MRI, CT scan, and/or PET/CT scan to check the status of the disease.

At the end of the study, the supporter Bristol-Myers Squibb Company will not continue to supply the study drugs, unless the study is extended. Your doctor will make sure that you receive appropriate standard of care or other appropriate treatment for your condition. You and/or your insurance provider may be responsible for the cost of treatment needed after the study is over.

## **Other Information**

You should not have any vaccinations while you are taking ipilimumab.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. These side effects will vary from person to person. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You should discuss these with the study doctor. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Tell the study staff about any side effects you may have, even if you do not think they are related to the study drug/procedures.

Nivolumab, ipilimumab, and SBRT may cause low blood cell counts (red blood cells, platelets, and/or white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

### BMS-986156 side effects

This is an early study of BMS-986156, so the side effects are not well known. Based on early human studies, BMS-986156 may cause:

- swelling (arms/legs)
- fatigue
- headache

- abdominal pain
- nausea/vomiting
- loss of appetite
- diarrhea

- pain (including back pain)
- difficulty breathing
- worsening/growth of a tumor

### **Nivolumab Side Effects**

# Common (occurring in more than 20% of patients)

- fatigue/lack of energy
- headache
- fever
- skin rash
- itching
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- high blood levels of fat (possible heart disease and/or stroke)

- high blood sugar (possible diabetes)
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- abdominal pain
- diarrhea
- loss of appetite
- nausea
- constipation
- abnormal digestive blood test (possible inflammation of the pancreas)

- low blood cell counts (red, white, platelets)
- abnormal liver test (possible liver damage and/or yellowing of the skin and/or eyes)
- pain
- abnormal kidney test (possible kidney damage)
- weakness
- · difficulty breathing
- cough
- infection

# Occasional (occurring in 3-20% of patients)

- swelling (arm/leg)
- dizziness
- skin redness
- patches of skin color loss
- overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)
- inflammation of the thyroid gland (possible tenderness in the neck)
- vomiting
- inflammation of the intestines

- mouth blisters/sores (possibly difficulty swallowing)
- abnormal blood test (possible pancreas damage)
- nerve damage (possible numbness, pain, and/or loss of motor/sensory function)
- inflammation of nerves (possible pain and/or loss of motor or sensory function)

- joint disease
- build-up of fluid around the lungs
- lung inflammation (possible difficulty breathing)
- stuffy nose
- immune reaction (possible organ damage)
- immune system disease (possible dry mouth/eyes, fatigue, joint pain, and/or organ failure)

| • | hole in the intestines |
|-------------------------|------------------------|
| (possibly leaking conte | |
| | into the abdomen) |

- peripheral nerve palsy (weakness, numbness, tingling)
- muscle damage causing weakness
- infusion reaction (possible chills and/or hives)

If you have a stem cell transplant from a donor before or after you receive nivolumab, you may have an increased risk of complications, such as severe graft-versus-host disease (when transplanted donor tissue attacks the recipient's organs such as skin, liver, and/or intestines) and/or clotting of blood within the liver. Deaths have been reported in patients who received stem cell transplant from a donor before or after nivolumab therapy. If you decide to receive a stem cell transplant from a donor, please tell your transplant doctor that you received nivolumab in the past.

# Rare but serious (occurring in fewer than 3% of patients)

- blood vessel inflammation (possible bleeding and/or bruising)
- heart inflammation
- brain inflammation (possible paralysis and/or coma)
- damage to the nervous system (causing numbness and/or paralysis)
- paralysis of the nerves controlling the head and neck
- skin blisters
- diabetes requiring insulin
- severe high blood sugar due to uncontrolled diabetes

- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- inflammation of the pancreas (possible abdominal pain)
- liver damage (possibly due to blood clots)
- paralysis (face)
- uncontrolled movements
- inflammation inside the eye (possible vision problems)
- kidney failure
- breakdown of muscle tissue (possibly kidney failure)

- blockage in the lung (possible pain and/or shortness of breath)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- Vogt Koyanagi Harada syndrome -- pigmented tissue (possible eye pain/swelling, hearing loss, and/or loss of skin color)

# Frequency unknown

- migraine
- very severe blistering skin disease (loss of large portion of skin and/or
- hand-foot syndrome (palms of hands/soles of feet having pain, swelling, and blistering)
- weight loss

| ulcers of the skin and |
|------------------------|
| digestive tract) |

You may need to take drugs to reduce inflammation while taking nivolumab. Long-term use of these drugs may increase your risk of infection. These infections may occur anywhere and may be fatal. Treatment with antibiotic or antifungal drugs may be required to treat these infections.

The study drug works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

Nivolumab may cause serious side effects that affect your immune system. Some of these side effects start as inflammation in different areas of the body like the skin, hormone glands, pancreas, or appendix. Tell the study staff right away if you have diarrhea, nausea, vomiting, blurred vision, dizziness, fainting, or you are feeling cold all the time.

If you had an organ transplant, nivolumab may increase your risk for the transplant to be rejected by your body.

# **Ipilimumab Side Effects**

# Common (occurring in more than 20% of patients)

- fatigue
- headache
- itching and/or skin rash
- weight loss
- nausea
- diarrhea

- loss of appetite
- vomiting
- abnormal digestive blood test (possible inflammation of the pancreas)
- constipation
- low red blood cell counts
- abnormal liver tests (possible liver damage)

# Occasional (occurring in 3-20% of patients)

- fever
- difficulty sleeping
- death of skin tissue and skin sores
- very severe blistering skin disease (with loss of large portion of skin)
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- skin rash with blisters or bleeding
- pituitary gland failure (possible endocrine gland abnormality)
- abdominal pain
- inflammation of the intestines
- abnormal blood test (possible pancreas damage)
- abnormal liver tests (possible yellowing of the skin and/or eyes)
- liver damage
- abnormal kidney test (possible kidney damage)
- cough
- difficulty breathing

# Rare but serious (occurring in fewer than 3% of patients)

- blood vessel disease
- blood vessel inflammation (possible bleeding and/or bruising)
- leakage of fluids from blood vessels into surrounding tissue (possible difficulty breathing)
- heart inflammation
- inflammation of the tissue around the heart (possible chest pain)
- brain inflammation (possible paralysis and/or coma)
- immune system damage to the nervous system (causing numbness and/or paralysis)
- immune response (causing muscle weakness)
- nerve damage (loss of motor or sensory function)
- Cushing's syndrome (possible weakness, diabetes, and/or bone weakness)
- red, dry, scaly patches of thickened skin (psoriasis)

- skin rash (possible fever/lymph node swelling/inflammation of internal organs/abnormal blood cell counts)
- allergic skin reaction
- inflammation of the thyroid gland (possible tenderness in the neck)
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)
- overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- hole in the intestines (possibly leaking contents into the abdomen)
- inflammation of the pancreas (possible abdominal pain)
- stomach and/or small intestine ulcer

- anemia due to destruction of red blood cells
- bone marrow failure due to abnormal tissue growth
- liver failure
- liver damage due to inflammation
- muscle inflammation and weakness
- inflammation inside the eye (possible vision problems)
- partial hearing loss
- · kidney failure
- bronchiolitis obliterans (damage of the small airways with difficulty breathing)
- lung inflammation (possible difficulty breathing)
- multi-organ disease causing lesions, most often in the lungs (sarcoidosis)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- immune response
- infection

Ipilimumab may cause dehydration that may be severe enough to require hospitalization.

Ipilimumab may cause an increased risk of infection, such as pneumonia. This infection may occur anywhere (such as the brain/spinal cord, lungs, and/or blood). It may become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

Ipilimumab works by boosting the immune system. This may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

### **Radiation Therapy Side Effects**

It is not known how often the side effects of radiation therapy may occur.

| • swelling | skin changes (possible) | • nausea |
|---|---|---|
| <ul> <li>swelling of the arms or</li> </ul> | dryness, itching, | <ul><li>vomiting</li></ul> |
| torso | peeling, and/or | <ul><li>diarrhea</li></ul> |
| | blistering) | joint problems |
| | <ul> <li>hair loss at the</li> </ul> | <ul> <li>secondary cancers</li> </ul> |
| | treatment site | |
| | <ul><li>trouble swallowing</li></ul> | |

Radiation therapy may cause you to develop another type of cancer. Side effects may not occur for up to 6 months after radiation therapy is over. Side effects will vary depending on what part of the body is receiving radiation therapy.

**Using the study drugs together with SBRT** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

# Other Risks

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

The type of **genetic testing** being performed in this study will not provide you or your doctor information about diseases that are passed down in families. It will not tell the study researchers anything that will prevent you from getting health insurance, and it will not tell the study researchers anything about any diseases or conditions you may get in the future.

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active.

Birth Control Specifications: If you can become pregnant, you must use at least 1 acceptable form of birth control while you are on study and for 160 days after your last study treatment. Acceptable forms include:

- Implantable progestogen-only hormonal birth control that stops ovulation
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion ("tubes tied")
- Vasectomized partner

If you can father a child, you must use a condom while on study (even if you have had a vasectomy or if your partner is pregnant or breastfeeding) and for 220 days after your last treatment. Your female partner should use effective methods of birth control while you are on study and for 160 days after then your last treatment.

Males: Do not donate sperm while on study. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy.

Females: If you are pregnant, you will not be enrolled on this study.

Getting pregnant will result in your removal from this study.

### OPTIONAL PROCEDURES FOR THE STUDY

**Optional Procedure #1:** If you agree, leftover tumor tissue and blood will be stored in a research bank at MD Anderson for use in future research related to cancer.

Before your samples can be used for research, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson. The IRB is a committee of doctors, researchers, and community members. The IRB is responsible for protecting study participants and making sure all research is safe and ethical.

Your samples will be given a code number. No identifying information will be directly linked to your samples. Only the researcher in charge of the bank will have access to the code numbers and be able to link the samples to you. This is to allow medical data related to the samples to be updated as needed.

There are no benefits to you for taking part in the optional procedures. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

### **Optional Procedure Risks:**

MD Anderson and others can learn about cancer and other diseases from your **banked samples**. In the future, people who may do research with these samples may need to know more information about your health. This information may be collected

from your medical record. MD Anderson will make reasonable efforts to preserve your privacy, but cannot guarantee complete privacy. Sometimes your samples may be used for genetic research about diseases that are passed on in families.

The type of **genetic testing** being performed in this study will not provide you or your doctor information about diseases that are passed down in families. It will not tell the study researchers anything that will prevent you from getting health insurance, and it will not tell the study researchers anything about any diseases or conditions you may get in the future.

If you withdraw your consent to the storage of leftover samples in the tissue bank, then they will no longer be collected for storage. Any of your samples that remain in the tissue bank will no longer be used for research and will be destroyed.

However, if any of your de-identified samples were already released for research purposes before you withdrew consent, MD Anderson will not be able to destroy them.

### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to allow leftover tumor tissue to be collected and stored in a research bank at MD Anderson for use in future research related to cancer?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or Bristol-Myers Squibb for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary

manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Joe Y. Chang, at 713-563-2300) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, Bristol-Myers Squibb, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is supported by: Bristol-Myers Squibb.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

### **Future Research**

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data and/or samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or samples are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### Genetic Research

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment.

### **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Bristol-Myers Squibb, who is a supporter of this study, and/or any future supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

Bristol-Myers Squibb is the supporter of this study and is providing the funding and drug support for this study. The samples will be stored in Dr. Chang's laboratory at MD Anderson. The following individuals will have access to this location: Maria Angelica Cortez, Hampartsoum Barsoumian, and Fatemeh Masrorpour.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT **LEGALLY AUTHORIZED REPRESENTATIVE (LAR)** The following signature line should only be filled out when the participant does not have the capacity to legally consent to take part in the study and/or sign this document on his or her own behalf SIGNATURE OF LAR DATE PRINTED NAME and RELATIONSHIP TO PARTICIPANT <u>WITNESS TO CONSENT</u> I was present during the explanation of the research to be performed under Protocol 2018-0419. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE

PRESENTATION (OTHER THAN PHYSICIAN OR STUDY

CHAIR)

| A witness signature is only required for vulnerable adult participants. If witnessing the assen pediatric participant, leave this line blank and sign on the witness to assent page instead. | t of a |
|---|---|
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her autrepresentative, using language that is understandable and appropriate. I bel have fully informed this participant of the nature of this study and its possible and risks and that the participant understood this explanation. | ieve that I |
| PERSON OBTAINING CONSENT D. | ATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT TRANSLATOR I have translated the above informed consent as written (without additions or subtractions) into and assisted the peop (Name of Language) obtaining and providing consent by translating all questions and responses d consent process for this participant. | le |
| NAME OF TRANSLATOR SIGNATURE OF TRANSLATOR DAT | E |
| ☐ Please check here if the translator was a member of the research team. checked, a witness, other than the translator, must sign the witness line below | • |
| SIGNATURE OF WITNESS TO THE VERBAL TRANSLATION (OTHER THAN TRANSLATOR, PARENT/GUARDIAN, OR STUDY CHAIR) | ATE |

PRINTED NAME OF WITNESS TO THE VERBAL TRANSLATION